CLINICAL TRIAL: NCT05288933
Title: Instrument-Assisted Soft Tissue Mobilization Versus High Power Pain Threshold Ultrasound In Management Of Upper Trapezius Myofascial Trigger Points: Randomized Controlled Trial
Brief Title: Instrument-Assisted Soft Tissue Mobilization Versus High Power Pain Threshold Ultrasound For Trapezius Myofascial Trigger Points
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Kamel Ibrahim El sayed, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003544
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Myofascial Pain Syndrome of Neck
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (A) conventional physical therapy (Active Comparator): 20 participants will receive conventional physical therapy.TENS, the frequency of the current is 100 Hz and the duty cycle is 250 microseconds, three times per week for 4 weeks. Ultrasound waves, frequency 1 MHz with intensity 1 W/cm2, a pulsed mode for 5 minutes, three times per week for 4 weeks, passive stretching, and isometric exercises three times per week for 4 weeks.
  Interventions: Device: Instrument assisted soft tissue mobilization ( IASTM ) and Ultrasound
- Group (B )IASTM and conventional physical therapy (Experimental): 20 participants will receive Instrument-Assisted Soft Tissue Mobilization (IASTM) and conventional physical therapy, the M2T blade will be used to find the exact areas of restriction in the upper trapezius. Then the M2T blade will be used, at an angle of 45 and using treatment planes 1, 2, and 3, to apply slow strokes along with the muscle, without causing any discomfort or pain, from the muscle origin to its insertion (sweeping technique), for approximately 3 min. This procedure will be repeated twice a week for four weeks
  Interventions: Device: Instrument assisted soft tissue mobilization ( IASTM ) and Ultrasound
- Group (C) HPPT US and conventional physical therapy (Experimental): 20 participants will receive High Power Pain Threshold Ultrasound (HPPT US) and conventional physical therapy. For the HPPT US, ultrasound waves will be applied to trigger points of the upper trapezius in continuous mode, and the power of ultrasound will first increase to the threshold pain level at intensity (1.5-2 W/cm) according to the patient for 4-5 seconds with the probe placed directly on the trigger point and held motionlessly and then reduced to one-half of that intensity for15 seconds with the probe placed directly on the trigger point and move in a circular motion and repeat this three times. This procedure will be repeated twice a week for two weeks
  Interventions: Device: Instrument assisted soft tissue mobilization ( IASTM ) and Ultrasound

INTERVENTIONS:
Device: Instrument assisted soft tissue mobilization ( IASTM ) and Ultrasound — Instrument-assisted soft tissue mobilization (IASTM) is a popular treatment for the myofascial limitation that is based on James Cyriax's rationale.
  High-power pain threshold ultrasound is a noninvasive approach used in myofascial pain syndrome ( MPS) treatment, and it has no serious adverse effects.
  Other Names: Ultrasound

SUMMARY:
the purpose of this trial is to compare the effectiveness of instrument-assisted soft tissue mobilization and high power pain threshold ultrasound on pain intensity, pressure pain threshold (PPT), neck range of motion, and neck function in participants with upper trapezius myofascial trigger points.

DETAILED DESCRIPTION:
Myofascial trigger points (MTPs) are hyperirritable, palpable nodules that form along with taut bands of muscle fibers. The trapezius is the muscle that is most commonly affected. MTPs can have a considerable impact on a person's daily activities and ability to work. Stretching exercises, ultrasound, massage, kinesiology taping, trigger point release, dry needling, laser, ischemic compression treatment, and high-power pain threshold ultrasound can all be used in a physical therapy program for myofascial pain and trigger points. There were previous studies on the effect of instrument-assisted soft tissue mobilization (IASTM) on upper trapezius myofascial trigger points that have shown positive effects such as reduction in pain level, improved neck function, and range of motion, increased activity level, and increased pressure pain threshold. There have been previous studies on the effect of high-power pain threshold ultrasound on upper trapezius trigger points that have shown a reduction in pain level, increased activity level, and increased pressure pain threshold. However till now, there is no study comparing the therapeutic potential of HPPT US and IASTM on upper trapezius trigger points, This study is conducted to compare the effect of instrument-assisted soft tissue mobilization (IASTM) and high-power pain threshold ultrasound ( HPPT US ) on upper trapezius trigger points. : Sixty participants ranging in age from 25 to 40 years old, from both genders, were diagnosed with active MTPs in the upper fibers of the trapezius muscle bilaterally. Participants were randomly allocated to the following three groups using sealed envelopes. Group (A) 20 participants received conventional physical therapy. Group (B) 20 participants received IASTM and conventional physical therapy. Group (C) 20 participants received HPPT US and conventional physical therapy for two weeks, twice per week.

ELIGIBILITY:
Inclusion Criteria: Having at least 1 active trigger point in bilateral upper trapezius muscles We will use a recommended diagnostic criterion to find active MTrPs which is:

The presence of a palpable taut band in the skeletal muscle, The presence of a hypersensitive spot in the taut band, Local twitch response provoked by snapping palpation Production of referred pain pattern in response to the compression of tender spots Spontaneous presence of typically referred pain pattern.

* A duration of symptoms of 2-4 weeks.
* Age between 25 and 40 years.
* Having a normal neurological examination result.
* Not having any evidence of infection or inflammation in laboratory tests.

Exclusion Criteria:- Existence of cervical disc hernia, advanced cervical osteoarthritis, radiculopathy, or myelopathy.

* Having trigger point injection or physical therapy in the last 6 months.
* Having a rheumatologic disease, such as fibromyalgia, rheumatoid arthritis, and spondyloarthritis, or hormonal diseases, such as hypothyroidism, hyperthyroidism, or hyperparathyroidism.
* Existence of kyphosis, scoliosis, forward head posture, or cervical-genic headache.
* History of spine surgery.
* Having a cardiovascular problem

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-06-12 (Actual); Study Completion 2022-06-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity | four weeks
  Pain intensity will be measured by the Visual Analogue Scale (VAS). It consists of a horizontal or vertical line, usually 10 cm long. The extremes of the line are labeled as "no pain" and "worst pain"
  3-Neck Range of motion : by Cervical ROM 3- Neck function: by Arabic version of the Neck Disability
Pressure pain threshold (PPT) | four weeks
  Pressure pain threshold (PPT) will be measured by a Pressure Algometer.
Neck Range of motion | four weeks
  Neck Range of motion will be measured by Cervical ROM
Neck function | four weeks
  Neck function will be measured by the Arabic version of the Neck Disability Index (ANDI). A total score of 0-4 indicated no disability. A score of 5-14 indicated mild disability, a score of 15-24 indicated moderate disability, a score of 25-34 indicated severe disability, and a score of 35 or greater indicated complete disability

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt